CLINICAL TRIAL: NCT03832322
Title: Water Exchange Colonoscopy Decreased Adenoma Miss Rates in the Right and Proximal Colon: An Observational Study Using A Tandem Colonoscopy Approach
Brief Title: Adenoma Miss Rate With Water Exchange vs Carbon Dioxide Colonoscopy
Status: Completed | Type: Observational
Sponsor: Evergreen General Hospital, Taiwan (Other)
Responsible Party: Principal Investigator, Chi-Liang Cheng, M.D., Evergreen General Hospital, Taiwan
Other Study IDs: EGH-2018
Record Dates: First submitted 2019-02-02; First posted 2019-02-06 (Actual); Results first posted 2019-05-10 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Colonic Adenoma; Water Exchange Colonoscopy
Keywords: Adenoma miss rate; Adenoma detection rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Water exchange colonoscopy: During the insertion phase of the first-pass colonoscopy, water exchange (WE) method was used. WE entailed the infusion of water to open the lumen and sequentially suction of water. When the cecum was reached and after most of the water was suctioned to collapse the cecal lumen, CO2 was opened during the withdrawal phase of the first-pass colonoscopy. After the first complete withdrawal of the colonoscope, a second colonoscopic examination aided by CO2 insufflation during insertion and withdrawal was performed by the same endoscopist. The colonoscope was reinserted into the cecum as quickly as possible, and the entire colon was re-examined. Polyp resection was carried out during insertion and withdrawal of the first- and second-pass examinations.
  Interventions: Procedure: Water exchange colonoscopy; Procedure: CO2 insufflation colonoscopy
- CO2 insufflation colonoscopy: During the first-pass colonoscopy, the procedure was performed in the usual fashion, with minimal CO2 insufflation to aid insertion. Cleaning of colon was predominantly performed during withdrawal. After the first complete withdrawal of the colonoscope, a second colonoscopic examination aided by CO2 insufflation during insertion and withdrawal was performed by the same endoscopist. The colonoscope was reinserted into the cecum as quickly as possible, and the entire colon was re-examined. Polyp resection was carried out during insertion and withdrawal of the first- and second-pass examinations.
  Interventions: Procedure: CO2 insufflation colonoscopy

INTERVENTIONS:
Procedure: Water exchange colonoscopy — During back-to-back colonoscopy, the first examination was completed with water exchange during insertion and CO2 insufflation during withdrawal. The second examination was completed with CO2 insufflation during both the insertion and withdrawal.
  Groups: Water exchange colonoscopy
Procedure: CO2 insufflation colonoscopy — During back-to-back colonoscopy, the first examination was completed with CO2 insufflation during both the insertion and withdrawal. The second examination was also completed with CO2 insufflation during both the insertion and withdrawal.

SUMMARY:
This was an observational study comparing consecutive group of WE and CO2 insufflation in terms of right and proximal colon AMR by tandem colonoscopy.

DETAILED DESCRIPTION:
This was a prospective observational study to assess how WE colonoscopy would fit into clinical and research practices. We first observed whether optimal WE colonoscopy decreased the AMR in the right and proximal colon in a tandem approach. If WE did lower the AMR as compared with data in the literature, a randomized RCT deserves to be studied. For the calculation of sample size in the upcoming RCT, the AMR in the CO2 group would be collected. The differences of the AMRs in the right and proximal colon determined by tandem colonoscopy using WE or CO2 insufflation would then be compared.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients aged 20 years or older undergoing colonoscopy for screening and surveillance indications were considered for enrollment.

Exclusion Criteria:

* familial adenomatous polyposis and hereditary non-polyposis CRC syndrome, personal history of inflammatory bowel disease, previous colonic resection, inability to achieve cecal intubation, obstructive lesions of the colon, poor colon preparation, inability to completely remove a polyp, gastrointestinal bleeding, allergy to fentanyl or midazolam, American Society of Anesthesiology classification of physical status grade 3 or higher, mental retardation, pregnancy, and refusal to provide a written informed consent.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 86 eligible patients completed first-pass colonoscopy with WE insertion and CO2 withdrawal, followed by back-to-back second-pass colonoscopy with CO2 insertion and CO2 withdrawal during July 9 to Oct 12, 2018; Another 86 eligible patient completed first-pass colonoscopy with CO2 insertion and CO2 withdrawal, followed by back-to-back second-pass colonoscopy with CO2 insertion and CO2 withdrawal during Oct 15 to Nov 21, 2018.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Liang Cheng, Principal Investigator — Evergreen General Hospital, Taoyuan, Taiwan
Locations (1):
- Evergreen General Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Cheng CL, Kuo YL, Hsieh YH, Tang JH, Leung FW. Water exchange colonoscopy decreased adenoma miss rates compared with literature data and local data with CO2 insufflation: an observational study. BMC Gastroenterol. 2019 Aug 14;19(1):143. doi: 10.1186/s12876-019-1065-2. PMID 31412789

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Water Exchange Colonoscopy | CO2 Insufflation Colonoscopy
Started | 89 | 87
Completed | 86 | 86
Not Completed | 3 | 1
Not completed — Failed cecal intubation in 2nd exam | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Water Exchange Colonoscopy: During the insertion phase of the first-pass colonoscopy, WE method was used. When the cecum was reached, CO2 was opened during the withdrawal phase of the first-pass colonoscopy. After the first complete withdrawal of the colonoscope, a second colonoscopic examination aided by CO2 insufflation during insertion and withdrawal was performed by the same endoscopist. The colonoscope was reinserted into the cecum as quickly as possible, and the entire colon was re-examined. Polyp resection was carried out during insertion and withdrawal of the first- and second-pass examinations.
- Total: Total of all reporting groups
Arm/Group | Water Exchange Colonoscopy | CO2 Insufflation Colonoscopy | Total
Number analyzed (Participants) | 86 | 86 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (10.7) | 52.9 (9.6) | 53.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 39 | 82
  Male | 43 | 47 | 90
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Taiwan | 86 | 86 | 172

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Overall Detected Adenomas Missed During the First Right-Colon Colonoscopy
Description: Right-colon (cecum, A-colon, hepatic flexure) adenomas detected on the second-pass examination were used for the calculation of adenoma miss. Adenoma miss rate was calculated as the number of adenomas missed in the first colonoscopy divided by the total number of adenomas detected during both the first and second colonoscopies.
Time Frame: During procedure, approximately 1.5 hours
Measure: Mean (95% Confidence Interval); unit: percentage of detected adenomas
Arm/Group | CO2 Insufflation Colonoscopy | Water Exchange Colonoscopy
Number analyzed (Participants) | 86 | 86
percentage of detected adenomas | 33.8 [23.2 to 45.7] | 17.5 [9.1 to 29.1]

2. Primary Outcome: Percentage of Overall Detected Adenomas Missed During the First Proximal-Colon Colonoscopy
Description: Proximal-colon (cecum, A-colon, hepatic flexure, T-colon) adenomas detected on the second-pass examination were used for the calculation of adenoma miss. Adenoma miss rate was calculated as the number of adenomas missed in the first colonoscopy divided by the total number of adenomas detected during both the first and second colonoscopies.
Time Frame: During procedure, approximately 1.5 hours
Measure: Mean (95% Confidence Interval); unit: percentage of detected adenomas
Arm/Group | Water Exchange Colonoscopy | CO2 Insufflation Colonoscopy
Number analyzed (Participants) | 86 | 86
percentage of detected adenomas | 15.5 [8.5 to 25.0] | 30.4 [22.0 to 39.8]

ADVERSE EVENTS:
Time Frame: one month
Arm/Group | Water Exchange Colonoscopy | CO2 Insufflation Colonoscopy
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/86
Other Adverse Events (participants affected / at risk) | 0/86 | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/22/NCT03832322/Prot_SAP_002.pdf